CLINICAL TRIAL: NCT03750487
Title: Home Visitation Enhancing Linkages Project (HELP 2.0)
Brief Title: Home Visitation Enhancing Linkages Project
Acronym: HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HELP 2.0; R34DA045831 (NIH)
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-screening & brief intervention (e-SBI) (Experimental): A two-session (20 minutes each) computer-delivered screening and brief motivational intervention targeting alcohol and drug use. Computerized screening is conducted using the ASSIST. Session 1 of the BI includes personalized feedback, readiness to change interventions, and goal setting around substance use. Session 2 will contain motivational content reinforcing engagement in home visiting and information around other challenges mothers may experience including tobacco use, postpartum depression, and intimate partner violence.
  Interventions: Behavioral: e-screening & brief intervention (e-SBI)
- Control (Sham Comparator): The control group will receive a similar 2-session brief motivational intervention. Session 1 focuses on nutrition and healthy eating, session 2 focuses on exercising while pregnant or in the postpartum period.
  Interventions: Behavioral: Control e-SBI

INTERVENTIONS:
Behavioral: e-screening & brief intervention (e-SBI) — Computer-delivered screening and brief motivational intervention targeting alcohol and drug use + goal-setting and content reinforcement
  Arms: e-screening & brief intervention (e-SBI)
Behavioral: Control e-SBI — Computer-delivered screening and brief motivational intervention targeting healthy eating and exercise
  Arms: Control

SUMMARY:
A small pilot randomized controlled trial (RCT) will be conducted to test the impact of an electronic screening and brief intervention (e-SBI) on reduction in substance use (measured via self-report), associated symptoms (depression and parenting stress), and improvement in home visiting retention and substance use treatment engagement. While a pilot RCT was originally planned, the study experienced significant delays and recruitment challenges due to the COVID-19 pandemic. Therefore, after review by the DSMB and study sponsor, the decision was made to eliminate the randomization and assign all participants to the intervention condition to evaluate feasibility and acceptability of the intervention.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to pilot test an electronic screening and brief intervention (e-SBI) that will be adapted for use with pregnant and postpartum women in home visiting (HV) programs. The e-SBI will be tested in a small randomized trial in two home visiting sites, with 20 home visitors and 40 clients. Home visitors will be randomized to the control intervention or the e-SBI. Clients will be surveyed at baseline, and 3- and 6- month follow-up to track e-SBI impacts on reduction in substance use (measured via self-report), associated symptoms (depression and parenting stress), and improvement in home visiting retention and substance use treatment engagement.

While a pilot RCT was originally planned, the study experienced significant delays and recruitment challenges due to the COVID-19 pandemic. Therefore, after review by the DSMB and study sponsor, the decision was made to eliminate the randomization and assign all participants to the intervention condition to evaluate feasibility and acceptability of the intervention. Total enrollment was N = 14. Four participants were assigned to the control condition prior to elimination of randomization. The remaining 10 participants were assigned to the intervention condition. Primary study outcomes were feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking,
* 18 years or older,
* pregnant or up to 3 months postpartum,
* newly enrolling in home visiting with a participating home visitor,
* not currently attending substance use treatment

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Dauber, PhD, Principal Investigator — Partnership to End Addiction (formerly CASAColumbia)
Locations (1):
- Partnership to End Addiction - 485, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-screening & Brief Intervention (e-SBI) | Control
Started | 10 | 4
Completed | 10 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-screening & Brief Intervention (e-SBI) | Control | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (4.5) | 30.4 (3.4) | 27.2 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 0 | 2 | 2
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 7 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: e-SBI Session 1 Completion Rate
Description: e-SBI session 1 completion rate (% of participants who completed e-SBI session 1)
Time Frame: Upon completion of e-SBI session 1, approximately 2-4 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | E-screening & Brief Intervention (e-SBI) | Control
Number analyzed (Participants) | 10 | 4
Participants
  Completed e-SBI session 1 | 8 | 4
  Did not complete e-SBI session 1 | 2 | 0

2. Primary Outcome: Acceptability: Satisfaction With e-SBI Session 1 (Intervention Group Only)
Description: 8-item user satisfaction survey based on the Technology Acceptance Model completed after each e-SBI session.
  The scale was developed by Ondersma in prior studies of the e-SBI, it does not have a formal title. The scale measures satisfaction with the e-SBI session.
  The following items are included in the scale:
  1. How much did you like this session?
  2. How easy was it to use this program?
  3. How interesting was this session?
  4. How respectful was this session?
  5. How much were you bothered by parts of this session? (reverse scored)
  6. How much did this session get you thinking about your substance use?
  7. How much did you feel you were helped during this session?
  8. How interested are you in working with the program again? Items were rated on a 1 to 5 Likert scale. Average across all 7 items was calculated, with item 5 reverse scored. Possible range of scores is 1 to 5. Higher scores indicate higher satisfaction with the e-SBI session.
Time Frame: Upon completion of e-SBI session 1, approximately 2-4 weeks after enrollment
Population: Only 4 people completed the acceptability scale following e-SBI session 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E-screening & Brief Intervention (e-SBI)
Number analyzed (Participants) | 4
units on a scale | 4.03 (.45)

3. Primary Outcome: Feasibility: e-SBI Session 2 Completion Rate
Description: e-SBI session 2 completion rate (% of participants who completed e-SBI session 2)
Time Frame: Upon completion of e-SBI session 2 (approximately 4-6 weeks after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | E-screening & Brief Intervention (e-SBI) | Control
Number analyzed (Participants) | 10 | 4
Participants
  Completed e-SBI session 2 | 7 | 4
  Did not complete e-SBI session 2 | 3 | 0

4. Primary Outcome: Acceptability: Satisfaction With e-SBI Session 2 (Intervention Group Only)
Description: as for outcome 2
Time Frame: Upon completion of e-SBI session 2, approximately 4-6 weeks after enrollment
Population: 7 people completed the acceptability scale following e-SBI session 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E-screening & Brief Intervention (e-SBI)
Number analyzed (Participants) | 7
units on a scale | 3.93 (.31)

ADVERSE EVENTS:
Time Frame: Approximately 6 weeks (time from enrollment until completion of e-SBI sessions).
Description: Adverse events: any untoward medical occurrence that occurs during administration of an intervention, which may or may not have a causal relation with the intervention.
  Serious adverse events: any medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; creates persistent or significant disability/incapacity, or a congenital anomaly/birth defects.
Arm/Group | E-screening & Brief Intervention (e-SBI) | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 0/10 | 0/4

LIMITATIONS AND CAVEATS:
There were many delays and challenges associated with the COVID-19 pandemic. Due to disruptions in the home visiting service system caused by the pandemic, recruitment for the study was extremely slow. After enrolling the first 4 participants, we made the decision along with the DSMB, the IRB, and the funder to change the design from an RCT to a single-condition pre-post feasibility study, with all participants assigned to the intervention condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03750487/Prot_SAP_000.pdf